CLINICAL TRIAL: NCT00210223
Title: Radiofrequency of Breast Cancers : Pilot Study in Non Surgical Patients
Brief Title: Radiofrequency of Breast Cancers in Non Surgical Patients
Acronym: RF-SEIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB2004-16
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Radiofrequency; Percutaneous technique; breast cancer; tolerance
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: In this prospective, single-arm study, we aimed to determine the efficacy and patient tolerance of ultrasonography (US)-guided percutaneous RF ablation with endocrine therapy for elderly patients with breast cancer who decline or are not candidates for surgery

ARMS (1):
- US-RF + endocrine therapy (Experimental): ultrasonography (US)-guided percutaneous radiofrequency (RF) ablation with endocrine therapy
  Interventions: Procedure: ultrasonography (US)-guided percutaneous radiofrequency (RF) ablation with endocrine therapy

INTERVENTIONS:
Procedure: ultrasonography (US)-guided percutaneous radiofrequency (RF) ablation with endocrine therapy — ultrasonography (US)-guided percutaneous radiofrequency (RF) ablation with endocrine therapy

SUMMARY:
To determine the efficacy and tolerance of ultrasonography (US)-guided percutaneous radiofrequency (RF) ablation with endocrine therapy in elderly patients with breast cancer who decline or are not candidates for surgery.

DETAILED DESCRIPTION:
There is increasing demand for minimally invasive treatments for small breast malignancies. This is due in part to increased availability of improved treatment approaches, with the introduction of neoadjuvant strategies, and for cosmetic reasons. Moreover, with the introduction of breast cancer screening programs, tumors are frequently diagnosed earlier and at a smaller size, enabling breast-conserving treatment with lumpectomy followed by whole-breast radiation therapy. For elderly patients, however, various physiologic alterations, comorbid diseases, and higher risk of complications are often perceived as contraindications to breast-conserving methods). In addition, elderly cancer patients generally receive fewer surgeries than younger patients. In this context, radiofrequency (RF) ablation is emerging as a minimally invasive nonsurgical technique for the treatment of small breast malignancies. Several pilot studies have published RF ablation tolerance and feasibility results for patients of all ages with small breast cancers and for small cohorts of elderly patients, but there is a lack of prospective data on long-term follow- up and long-term efficacy for elderly patients. In this prospective, single-arm study, we aimed to determine the efficacy and patient tolerance of ultrasonography (US)-guided percutaneous RF ablation with endocrine therapy for elderly patients with breast cancer who decline or are not candidates for surgery.

ELIGIBILITY:
Inclusion criteria:

* Patients more than 70 years old
* Breast tumors with estrogen receptors
* Non surgical patients
* Life expectancy more than 6 months

Exclusion criteria:

* Presence of a pace maker
* Tumors measuring more than 30 mm on ultrasound evaluation, located less than 10 mm from skin, nipple, or pectoral muscle
* Coagulation disorders
* Contra indications to magnetic resonance imaging or computed tomography with contrast medium injection
* Non visible lesions on magnetic resonance imaging or computed tomography with contrast medium injection

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne VALENTIN, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié - Centre Régional de Luttre Contre le Cancer de Bordeaux et du Sud Ouest, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palussiere J, Henriques C, Mauriac L, Asad-Syed M, Valentin F, Brouste V, Mathoulin-Pelissier S, Tunon de Lara C, Debled M. Radiofrequency ablation as a substitute for surgery in elderly patients with nonresected breast cancer: pilot study with long-term outcomes. Radiology. 2012 Aug;264(2):597-605. doi: 10.1148/radiol.12111303. Epub 2012 Jun 12. PMID 22692040

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | US-RF + Endocrine Therapy
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | US-RF + Endocrine Therapy
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] | 79 [70 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease Recurrence One Year After the Intervention.
Description: The intervention was ultrasonography (US)-guided percutaneous radiofrequency (RF) ablation with endocrine therapy.
  Recurrence was assessed based on follow-up with dynamic contrast material-enhanced (DCE) magnetic resonance (MR) imaging).
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | US-RF + Endocrine Therapy
Number analyzed (Participants) | 21
Participants | 1

2. Secondary Outcome: Number of Participants With Disease Recurrence at 5 Years
Description: as for outcome 1
Time Frame: 5 years after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | US-RF + Endocrine Therapy
Number analyzed (Participants) | 21
Participants | 4

ADVERSE EVENTS:
Time Frame: 5 years
Description: Adverse events were not collected
Arm/Group | US-RF + Endocrine Therapy
All-Cause Mortality (participants affected / at risk) | 4/21
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes